CLINICAL TRIAL: NCT01982396
Title: Pharmacokinetic Study of Twice Daily vs Once Daily Lamivudine and Abacavir as Part of Combination Antiretroviral Therapy in Children With HIV Infection
Brief Title: Pharmacokinetic (PK) Study of Twice Daily vs Once Daily Lamivudine (3TC) and Abacavir (ABC) as Part of Combination Antiretroviral Therapy (ART) in HIV Infected Children
Acronym: PENTA 13
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PENTA 13
Record Dates: First submitted 2013-10-25; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infection
Keywords: HIV; paediatric; Abacavir; lamivudine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Twice daily (Active Comparator)
  Interventions: Drug: ABC Twice Daily; Drug: 3TC Twice Daily
- Once daily (Experimental)
  Interventions: Drug: ABC Once Daily; Drug: 3TC Once Daily

INTERVENTIONS:
Drug: ABC Twice Daily
  Arms: Twice daily
Drug: ABC Once Daily
  Arms: Once daily
Drug: 3TC Once Daily
  Arms: Once daily
Drug: 3TC Twice Daily
  Arms: Twice daily

SUMMARY:
Cross-over 28 week study of the plasma pharmacokinetic profiles of twice daily 3TC (4mg/kg/dose BD) with once daily 3TC (8mg/kg/dose OD) and twice daily ABC (8mg/kg/dose BD) with daily ABC (16mg/kg/dose OD) where one or both drugs are being taken as part of combination antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children with definitive HIV infection
* Age > 2 and < 13 years
* Currently on combination ART including 3TC and / or ABC, for at least 6 months, with stable CD4 cell count and HIV RNA viral load and expected to stay on this regimen for at least a further 3 months.

Exclusion Criteria:

* • Intercurrent illness

  * Receiving concomitant therapy except prophylaxis against Pneumocystis carinii pneumonia (PCP)
  * Abnormal renal or liver function (grade 3 or above)

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2003-01; Primary Completion 2004-02 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) of lamivudine after qd and bid dosing | week 0 and Week 4
Cmin of lamivudine after qd and bid dosing | week 0 and week 4
Cmax of lamivudine after qd and bid dosing | week 0 and week 4
AUC of abacavir after qd and bid dosing | week 0 and week 4
Cmin of abacavir after qd and bid dosing | week 0 and week 4
Cmax of abacavir after qd and bid dosing | week 0 and week 4

SECONDARY OUTCOMES:
To describe trough intracellular levels of 3TC on twice daily and once daily dosage regimens | Week 0 and week 4

OTHER OUTCOMES:
To describe patient and family acceptability of and adherence to once daily compared to twice daily dosing | week -2 and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Vas Novelli, MD, Principal Investigator — Great Ormond Street Hospital for Children, London, UK; Hermione Lyall, MD, Principal Investigator — St. Mary's Hospital, London, UK
Locations (2):
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - St. Mary's Hospital, London

REFERENCES:
- [Background] Bergshoeff A, Burger D, Verweij C, Farrelly L, Flynn J, Le Prevost M, Walker S, Novelli V, Lyall H, Khoo S, Gibb D; PENTA-13 Study Group. Plasma pharmacokinetics of once- versus twice-daily lamivudine and abacavir: simplification of combination treatment in HIV-1-infected children (PENTA-13). Antivir Ther. 2005;10(2):239-46. PMID 15865218
- [Background] LePrevost M, Green H, Flynn J, Head S, Clapson M, Lyall H, Novelli V, Farrelly L, Walker AS, Burger DM, Gibb DM; Pediatric European Network for the Treatment of AIDS 13 Study Group. Adherence and acceptability of once daily Lamivudine and abacavir in human immunodeficiency virus type-1 infected children. Pediatr Infect Dis J. 2006 Jun;25(6):533-7. doi: 10.1097/01.inf.0000222415.40563.d4. PMID 16732152
- See also: PENTA 13 publications and presentations — http://www.penta-id.org/hiv/penta-trials/penta-trials-publications/49-penta-13.html